CLINICAL TRIAL: NCT06952608
Title: The Effect of Ciprofol on Intraoperative Hypotension in Elderly Patients Receiving Renin-angiotensin System Inhibitors: a Prospective, Randomized Controlled Trial
Brief Title: Effect of Ciprofol on Intraoperative Hypotension in Elderly Patients Receiving Renin-angiotensin System Inhibitors
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2025-0279
Record Dates: First submitted 2025-04-13; First posted 2025-05-01 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-04

CONDITIONS: Intraoperative Hypotension; Ciprofol; Renin-angiotensin System Inhibitors

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ciprofol Group (Experimental): General anesthesia induction and maintenance were performed using ciprofol.
  Interventions: Drug: Ciprofol group
- Propofol group (Placebo Comparator): General anesthesia induction and maintenance were performed using propofol.
  Interventions: Drug: Propofol group

INTERVENTIONS:
Drug: Ciprofol group — General anesthesia induction and maintenance were performed using ciprofol.
  Arms: Ciprofol Group
Drug: Propofol group — General anesthesia induction and maintenance were performed using propofol.
  Arms: Propofol group

SUMMARY:
The prevention of intraoperative hypotension could reduce postoperative organ injury and mortality, particularly in elderly patients receiving long-term renin-angiotensin system inhibitors. Previous meta-analyses suggest that ciprofol, a novel intravenous anesthetic agent, may provide improved hemodynamic stability compared to propofol; however, its precise effects on perioperative hemodynamics remain unclear. The study will assess whether ciprofol improves perioperative hemodynamic stability in elderly patients receiving renin-angiotensin system inhibitors.

DETAILED DESCRIPTION:
Elderly patients receiving long-term renin-angiotensin system inhibitors commonly exhibit reduced vascular elasticity, impaired cardiovascular reserve, and diminished compensatory mechanisms. Regular use of renin-angiotensin system inhibitors has thus emerged as a significant risk factor for intraoperative hypotension, increasing the potential for end-organ injury and closely correlating with postoperative complications such as myocardial injury, acute kidney injury, and increased mortality.

Ciprofol (HSK3486) is a novel intravenous anesthetic agent that has demonstrated efficacy non-inferior to propofol for induction and maintenance of general anesthesia, with an improved safety profile and fewer adverse effects. Recent meta-analyses indicate that ciprofol administration is associated with a significantly reduced incidence of intraoperative hypotension compared with propofol; however, robust evidence from randomized controlled trials (RCTs) remains limited. The present study aims to evaluate the impact of ciprofol on perioperative hemodynamics in elderly patients receiving renin-angiotensin system inhibitors. Given the increased risk of intraoperative hypotension in this patient cohort, the investigation of hemodynamic stability with ciprofol holds substantial clinical significance and may inform anesthetic management strategies for this vulnerable population.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing elective abdominal surgery under general anesthesia
2. Duration of surgery exceeding 2 hours
3. Patients receiving long-term renin-angiotensin system inhibitor therapy (>3 months prior to surgery)
4. Age ≥ 65 years
5. ASA classification II-III
6. Informed consent was obtained from patients or their guardians

Exclusion Criteria:

1. History of allergy to opioids, propofol, or ciprofol components.
2. Anticipated difficult airway (limited mouth opening, restricted neck movement, or modified Mallampati grade III-IV) or difficult mask ventilation.

   Body mass index ≤18 or ≥35 kg/m².
3. Severe hepatic dysfunction (total bilirubin ≥3.0 mg/dL or AST/ALT ≥2 times the upper limit of normal).
4. Severe renal impairment (creatinine clearance ≤30 mL/min).
5. Cardiac diseases (AV block higher than first-degree, heart rate <50 bpm, severe arrhythmias, severe valvular heart disease, heart failure, or unstable angina on the day of surgery).
6. Preoperative cognitive impairment, cerebrovascular disease, or history of psychiatric illness.
7. Abnormal thyroid-stimulating hormone levels or history of thyroid replacement therapy.
8. Unstable asthma or history of asthma.
9. Alcohol abuse, drug abuse, chronic opioid dependence, or analgesic use exceeding 3 months.
10. Lactating or pregnant women.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2026-02-10 (Estimated); Study Completion 2026-04-10 (Estimated)

PRIMARY OUTCOMES:
The time-weighted average of hypotension | From the beginning to the end of the surgery
  The time-weighted average is measured by calculating the area under the threshold (AUT) divided by the total duration of surgery

SECONDARY OUTCOMES:
Time-weighted average of hypotension | within 15 minutes after induction of anesthesia
  The time-weighted average is measured by calculating the area under the threshold (AUT) divided by the total duration of induction.
Incidence of intraoperative hypotension | From the beginning to the end of the surgery
Dosage of vasoactive drugs | From the beginning to the end of the surgery
Success rate of general anesthesia induction | From the beginning to the end of the surgery
  MOAA/S score of 1 or less after administration of ciprofol or propofol, 1 or fewer top-up doses, and no use of rescue drug
Proportion of intraoperative time with BIS ≤ 60 | From the beginning to the end of the surgery
Total dosage of ciprofol and propofol | From the beginning to the end of the surgery
Total dosage of rescue drugs | From start of drug administration to MOAA/S ≤1 (up to 5 minutes)
Time to extubation | Perioperative
Incidence of intraoperative adverse events | From the beginning to the end of the surgery
Incidence of adverse events in the PACU | during the PACU stay
Incidence of perioperative major adverse cardiovascular and cerebrovascular events | Periprocedural
Changes in Stroke Volume Variation (SVV) | Intraoperative
  Nomal value:≤10%,and higher scores mean a worse outcome.
Changes in Cardiac Index (CI) | Intraoperative
  Nomal value:2.5-4.0 L/min/m²,and values outside the normal range suggest worse clinical outcomes
Changes in Systemic Vascular Resistance Index (SVRI) | Intraoperative
  Nomal value :1970-2390 dyn·s·cm-⁵·m²,and values outside the normal range suggest worse clinical outcomes
Changes in Cerebral Oxygen Saturation (rSO₂) | Intraoperative
Postoperative complications | From enrollment to the end of treatment at 3 months
  delirium, myocardial injury, stroke, acute kidney injury, infection, sepsis, etc.

OTHER OUTCOMES:
Quality of Recovery-15 (QoR-15) score | 3 day after surgery
emergency delirium | Periprocedural
  RASS&CAM-ICU, delirium was judged according to whether there were positive features in the questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Min Yan, Study Director — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- The Second Affiliated Hospital of Zhejiang University anesthesiology department, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No